CLINICAL TRIAL: NCT06752603
Title: A Phase IIa, Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-center Trial to Evaluate the Efficacy and Safety of ONO-1110 in Patients With Hunner Type Interstitial Cystitis
Brief Title: A Clinical Study of ONO-1110 in Patients With Hunner Type Interstitial Cystitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-1110-06; jRCT2031240558 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hunner Type Interstitial Cystitis
Keywords: ONO-1110; ONO-1110-06; Hunner Type Interstitial Cystitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-1110 (Experimental): ONO-1110 tablets once a day
  Interventions: Drug: ONO-1110
- Placebo (Placebo Comparator): Placebo tablets once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-1110 — ONO-1110 tablets once a day
  Arms: ONO-1110
Drug: Placebo — Placebo tablets once daily
  Arms: Placebo

SUMMARY:
To Evaluate the Efficacy and Safety of ONO-1110 in Patients with Hunner Type Interstitial Cystitis

ELIGIBILITY:
Inclusion Criteria:

* Japanese (both sexes)
* Age (at the time of informed consent): 18 years and older
* Outpatient
* Patients who are considered capable of understanding the study procedures and completing the pain diary, bladder diary, and questionnaires appropriately by the investigator (sub-investigator）
* Patients given a diagnosis of HIC by cystoscopy
* Patients with chronic pelvic pain involving the bladder and lower urinary tract symptoms such as increased micturition and pollakiuria

Exclusion Criteria:

* Patients with a history and presence of chemical cystitis
* Patients with a history of bladder augmentation or radical cystectomy
* Patients with pain other than HIC that may affect assessments in this study
* Patients with a past history of or concurrent neurologic diseases that may affect assessments in this study
* Patients receiving medications for psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in weekly mean of average pain score from baseline to Week 12 of the treatment period | Up to 20 weeks
Adverse events | Up to 20 weeks

SECONDARY OUTCOMES:
Change in weekly mean of average pain score from baseline in each week | Up to 20 weeks
30%- and 50%-responder rates based on the weekly mean of average pain score | Up to 20 weeks
  proportions of participants whose weekly mean of average pain score has decreased by 30% and 50% from baseline, respectively
Change in weekly mean of worst pain score from baseline to each week | Up to 20 weeks
30%- and 50%-responder rates based on the weekly mean of worst pain score | Up to 20 weeks
  proportions of participants whose weekly mean of worst pain score has decreased by 30% and 50% from baseline, respectively
Change in Interstitial cystitis symptom index (ICSI) score from baseline | Up to 20 weeks
Change in Interstitial cystitis problem index (ICPI) score from baseline | Up to 20 weeks
Change in Average frequency of urination per day from baseline | Up to 20 weeks
Change in Frequency of nocturnal urination per day from baseline | Up to 20 weeks
Change in Mean volume voided per micturition in a day from baseline | Up to 20 weeks
Change in Maximum volume voided per micturition in a day from baseline | Up to 20 weeks
Change in Number of urgency episodes per day from baseline | Up to 20 weeks
Change in Patient Global Impression of Change (PGIC) score from baseline | Up to 20 weeks
Change in SF-12v2 score from baseline | Up to 20 weeks
Change in Hospital Anxiety and Depression Scale (HADS) score from baseline | Up to 20 weeks
Plasma ONO-1110 concentrations | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (20):
- Japan (20):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Harasanshin Hospital, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Japanese Red Cross Gifu Hospital, Gifu, Gifu
  - Kurosawa Hospital Health Park Clinic, Takasaki, Gunma
  - Niimura Hospital, Kagoshima, Kagoshima-ken
  - Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Rakuwakai Marutamachi Hospital, Kyoto, Kyoto
  - Ueda Clinic, Kyoto, Kyoto
  - Izumi Chuo Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto, Nagano
  - Nakamura Hospital, Beppu, Oita Prefecture
  - Okayama University Hospital, Okayama, Okayama-ken
  - Nanri Urological Clinic, Saga, Saga-ken
  - The Jikei University Hospital, Minato-Ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - The University Of Tokyo Hospital, Tokyo, Tokyo
  - Toyama Rosai Hospital, Uozu, Toyama
  - University Of Yamanashi Hospital, Chūō, Yamanashi
  - Nagasaki University Hospital, Nagasaki

IPD SHARING:
Plan to Share IPD: No